CLINICAL TRIAL: NCT01923610
Title: Safety and Immunological Response of a Boosting Dose of MVA-B in Healthy Volunteers After 4 Years of Receiving MVA-B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Juan A. Arnaiz, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RisVac02 boost
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: HIV Infections
Keywords: Low risk HIV infection; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Main (Experimental): MVA HIV-B
  Interventions: Biological: Experimental

INTERVENTIONS:
Biological: Experimental — Biological/Vaccine: MVA-B Modified Pox virus, strain MVA clade -B (expressing HIV-1 Bx08gp120 and IIIB gagpolnef)
  -~ 1 x 10e8 pfu/ml 3 immunisations at week 0, 4 and 16

SUMMARY:
24 healthy male and female volunteers who are at low risk of HIV infection and entered into the RISVAC02 study and were randomly allocated to receive 3 intramuscular injections of MVA-B at weeks 0, 4 and 16 will receive a boosting dose 4 years thereafter.

Participants will attend one of two clinical centres on at least 5 occasions over 16 weeks. These visits will comprise:

* Screening
* Trial entry and boosting immunisation
* Early follow-up after immunisation
* Follow-up x 2 including the final visit Participants will have blood and urine collected, and receive 1 immunisation. They will be counselled prior to and following a HIV test, and given health education on prevention of sexually transmitted infections including HIV. T

The two centres which participate are:

* Hospital Clinic, Barcelona and
* Hospital Gregorio Marañón, Madrid The primary objective is to explore the safety and immunogenicity of MVA-B.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* age between 18 and 55 years on the day of screening
* available for follow-up for the duration of the study (52 weeks from screening)
* able to give written informed consent
* at low risk of HIV and willing to remain so for the duration of the study low risk of HIV infection defined as: no history of injecting drug use in the previous ten years no gonorrhoea or syphilis in the last six months no high risk partner (e.g. injecting drug use, HIV positive partner) either currently or within the past six months no unprotected anal intercourse in the last six months no unprotected vaginal intercourse outside a relationship with a regular known/presumed HIV negative partner in the last six months
* willing to undergo a HIV test
* willing to undergo a genital infection screen
* if heterosexually active female, using an effective method of contraception with partner (combined oral contraceptive pill; injectable contraceptive; IUCD; consistent record with condoms if using these; physiological or anatomical sterility in self or partner) from 14 days prior to the first vaccination until 4 months after the last, and willing to undergo urine pregnancy tests prior to each vaccination
* if heterosexually active male, using an effective method of contraception with their partner from the first day of vaccination until 4 months after the last vaccination

Exclusion Criteria:

* positive for hepatitis B surface antigen, hepatitis C antibody, antibody responses to vaccinia or serology indicating active syphilis requiring treatment
* pregnant or lactating
* clinically relevant abnormality on history or examination including history of grand-mal epilepsy, severe eczema, immunodeficiency or use of immunosuppressives in preceding 3 months
* receipt of live attenuated vaccine within 60 days or other vaccine within 14 days of enrolment
* receipt of blood products or immunoglobin within 4 months of screening
* participation in another trial of a medicinal product, completed less than 30 days prior to enrolment
* history of severe local or general reaction to vaccination defined as local: extensive, indurated redness and swelling involving most of the front-lateral thigh or the major circumference of the arm, not resolving within 72 hours general: fever >= 39.5oC within 48 hours; anaphylaxis; bronchospasm; laryngeal
* HIV 1/2 positive or indeterminate on screening
* positive for hepatitis B surface antigen, hepatitis C antibody or serology indicating active syphilis requiring treatment
* grade 1 routine laboratory parameters
* unlikely to comply with protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Local adverse event | 12 weeks
  Grade 3 or above local adverse event (pain, cutaneous reactions including induration)
Grade 3 or above systemic adverse event | 12 weeks
  Grade 3 or above systemic adverse event (temperature, chills, headache, nausea, vomiting, malaise, and myalgia)
Grade 3 or above other clinical or laboratory adverse event | 12 weeks
  Grade 3 or above other clinical or laboratory adverse event confirmed at examination or on repeat testing respectively
Event attributable to vaccine leading to discontinuation | 12 weeks
  Any event attributable to vaccine leading to discontinuation of the immunisation regimen
Primary immunogenicity parameters | 12 weeks
  The primary immunogenicity parameters will be quantitative or present/absent, and are cellular responses - CD8/CD4+ T cell responses (ELISPOT) at week 2, 4 and 12 following the immunisations

SECONDARY OUTCOMES:
All grade 1 and 2 adverse events | 28 days of vaccination
Antibody responses | 12 weeks
  * binding titration to the construct MVAB
  * binding titration to and neutralisation of vaccinia
cellular responses | 12 weeks
  * CD8/CD4+ T cell responses (ELISPOT) at week 0
  * intracellular cytokine analysis at week 0, 2, 4 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Garcia, MD, Principal Investigator — Hospital Clínic i Provincial de Barcelona
Locations (2):
- Spain (2):
  - Hospital Clínic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital Universitario Gregorio Marañón, Madrid, Madrid

REFERENCES:
- [Derived] Guardo AC, Gomez CE, Diaz-Brito V, Pich J, Arnaiz JA, Perdiguero B, Garcia-Arriaza J, Gonzalez N, Sorzano COS, Jimenez L, Jimenez JL, Munoz-Fernandez MA, Gatell JM, Alcami J, Esteban M, Lopez Bernaldo de Quiros JC, Garcia F, Plana M; RISVAC02boost study. Safety and vaccine-induced HIV-1 immune responses in healthy volunteers following a late MVA-B boost 4 years after the last immunization. PLoS One. 2017 Oct 24;12(10):e0186602. doi: 10.1371/journal.pone.0186602. eCollection 2017. PMID 29065142